CLINICAL TRIAL: NCT00767559
Title: Prophylaxis Against Thromboembolic Disease Following Orthopaedic Surgeries on Extremities
Brief Title: Prophylaxis Against DVTs After Primary Hip and Knee Replacement Surgery
Acronym: DVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The New England Baptist Hospital (Other)
Responsible Party: Murray Bern, MD, New England Baptist Hostpital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEBH 2008-016
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Pulmonary Embolism
Keywords: Deep Vein Thrombosis, anticoagulants, surgery, pulmonary embolus, warfarin, fondaparinox
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis | interventions — Warfarin; Fondaparinux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Variable dose warfarin: 5 mg beginning the night before surgery, followed by 5mg the PM of surgery*, and then variable daily dose,until day 30 follow-up.
  (target INR 2.0-2.5)
  Interventions: Drug: warfarin
- 2 (Active Comparator): Fondaparinux:
  2.5 mg daily starting more than 6 hours following surgery and no later than 6 AM the next day*,or 6-8 hours after epidural catheter removal, and continued until follow-up (28 days +/-2) from day of surgery.
  Interventions: Drug: Fondaparinux:
- 3 (Active Comparator): Fixed Low Dose warfarin
  1 mg daily beginning 7 days preoperative, and continued at 1 mg daily follow-up at Day 28 (+/-2 days from surgery).
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: warfarin — 5 mg beginning the night before surgery, followed by 5 mg the PM of surgery*, and then variable daily dose, until day 28 (+/-2 days) from day of surgery follow-up. (target INR 2.0 -2.5)
  Other Names: Coumadin
  Arms: 1
Drug: Fondaparinux: — 2.5 mg daily starting more than 6 hours following surgery and no later than 6 AM the next day*, or 6-8 hours after epidural catheter removal, and continued until follow up day 28 (+/-2 days) from day of surgery.
  Other Names: Arixtra
  Arms: 2
Drug: warfarin — Fixed Low Dose warfarin
  1 mg daily beginning 7 days preoperative, and continued at 1 mg daily until follow-up 28 day (+/- 2 days) from day of surgery.
  Other Names: coumadin
  Arms: 3

SUMMARY:
The purpose of this research is to find a better way to prevent the post operative development of clots in the deep veins of the legs (also called Deep Vein Thrombosis or DVT). DVT causes redness, swelling, and pain in the involved leg(s). Long-term complications may include permanent swelling and pain of the leg(s), and even skin ulcers around the ankle. If clots form in a leg after surgery, and break off, they can move to the lungs and block the pulmonary artery (also called Pulmonary Emboli or PE). With PE there can be chest pain, chest tightness, shortness of breath, coughing up blood, heart failure, and occasionally death.

Doctors have studied ways to reduce these complications. These studies led to the development of drugs which interfere with your body's clotting processes. However, it is still unclear which drug and which drug schedule is best. This study will evaluate two of the standard FDA approved drugs using different dosing schedules.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Planned for elective primary arthroplasty for knee and hip disease at New England Baptist Hospital.
2. Over 20 years of age.
3. Normal baseline platelet count, prothrombin and partial thromboplastin times.
4. Signed consent.

Exclusion Criteria:

1. Surgery for acute fracture (< 4 weeks), septic joint, or extraction arthroplasty.
2. Patients with personal history of TED, or documented hypercoagulation disease.
3. Increased risk of hemorrhage, as from active gastric ulcer, or bleeding diathesis; or persistent intestinal or urinary tract bleed within the last year.

SPECIFIC AIMS:

This prospective, randomized study seeks to determine if there is an advantage for fixed, low dose of warfarin Thromboembolic Disease (TED) prophylaxis among patients undergoing elective lower extremity joint arthroplasty, as compared to variable dose warfarin and a low molecular weight heparin (LMWH). If confirmed as effective fixed, low dose warfarin would be an almost ideal prophylaxis against Deep Vein Thrombosis (DVT) and Pulmonary Embolus (PE): inexpensive, easy to administer, with minimal hemorrhagic potential, needing minimal laboratory support .

BACKGROUND AND SIGNIFICANCE:

A progression of studies has been performed to examine the efficacy of low dose warfarin. These studies demonstrated that low dose warfarin has antithrombotic activity, with little anticoagulant effect. Critical to this approach that the warfarin therapy be initiated prior to surgery. A summary of other studies offering supportive or conflicting data is available. (1-9)

1. Low dose warfarin (2mg) dampens activated coagulation. (1-3)
2. Two-step low dose warfarin begun 10-14 days pre-op is effective prophylaxis. (4)
3. Low dose warfarin (1mg) prevents DVT's surrounding central venous catheters when started 3 days before catheter insertion among patients at very high risk for subclavian DVT. (5,6)
4. Low dose warfarin (1mg) started 7 days prior to surgery is equal to variable dose warfarin for TED prophylaxis following hip arthroplasty. (7)
5. Low dose warfarin (1mg) started 7 days prior to surgery is effective TED prophylaxis for patients having hip replacement arthroplasties in retrospective study of 1003 patients. (8)

The sentinel study used a fixed low dose warfarin regimen given to patients at extreme risk for DVT. Patients requiring central venous catheters for chemotherapy for metastatic cancer participated in a randomized study of 0.0 mg vs.1.0 mg daily warfarin starting 3 days prior to catheter placement. Subclavian vein venograms were performed at the time of symptoms of subclavian vein DVT or after 90 days. When using this low dose warfarin schedule there was a reduction in the incidence of thrombosis from 37.5% to 9.5%. (p<0.05) Four patients acquired vitamin K-responsive prolongation of the PT due to concomitant advanced liver disease and/or malnutrition. Concentrations of factors II, VII, IX, X, and protein C showed no difference between treated and untreated patients. (5)

Two orthopedic surgery studies from NEBH on this question have been published. (7,8) The first was a pilot study of 100 patients demonstrated no difference between the effectiveness of low fixed dose and variable dose warfarin in a population of patients at high risk for TED (7) Patients studied were planning total hip replacement arthroplasty were randomized between the standard regimens using warfarin of 5 mg the night prior to surgery followed by variable dose (target PT 1.3 - 1.5 times normal) for 30-45 days, or the experimental regimen using 1 mg beginning 7 days prior to surgery and continued until follow up at 30-45 days. Ultrasounds of the deep veins of the legs were performed at baseline, at discharge following surgery, and at 30-45 day follow-up. There was no difference between the groups for incidence of venous thrombosis. The second study was a retrospective study of patients undergoing primary (833) or revision (170) hip replacement arthroplasty receiving 1 mg warfarin for 7 days before surgery, variable dose while in hospital, (INR target 1.5 - 2.0) followed by 1 mg daily until follow-up at 30-45 days. (8) Each patient used pneumatic followed by elastic compression stockings. Of these 1003 patients, with 9 lost to follow-up. Three patients had TED, including 1 PE and 2 DVT.

ELIGIBILITY:
Inclusion Criteria:

1. Planned for elective arthroplasty for knee and hip disease.
2. Over 20 years of age.
3. Normal baseline platelet count, prothrombin and partial thromboplastin times.
4. Signed consent.

Exclusion Criteria:

1. Surgery for acute fracture (< 4 weeks), septic joint, or extraction arthroplasty.
2. Patients with personal history of TED, or documented hypercoagulation disease.
3. Increased risk of hemorrhage, as from active gastric ulcer, or bleeding diathesis; or persistent intestinal or urinary tract bleed within the last year.
4. Hemorrhagic stroke; brain, spinal, or ophthalmologic surgery in previous 6 months.
5. Liver enzymes or bilirubin greater than 2 x normal.
6. Decreased renal function with GFR < 30ml/min. (24-27)
7. Cancer in last 1 year, other than localized cancers of the skin.
8. Requires chronic anticoagulation with warfarin or heparins.
9. Requires chronic platelet function suppressive therapy for coronary or peripheral artery stents..
10. Prior adverse reaction to any of the study drugs.
11. Pregnancy
12. Uncontrolled hypertension

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome based upon intent to treat: Composite outcome of | 28 days
Ultrasound or venogram confirmed deep vein thrombosis. | 28 days
Lung scan, pulmonary angiogram or CTA confirmed pulmonary embolus. | 28 days
Death due to TED | 28 days

SECONDARY OUTCOMES:
Patient compliance with preoperative and post-operative medication schedule. Not enough space to note all measures | 28 days
Distribution of proximal vs distal deep vein thrombosis of the leg | 28 days
Amount of intraoperative bleeding | follow until Dec. 31, 2010
Amount of postoperative bleeding A. transfusion requirement B. Hematomas requiring intervention, or other bleed clinically thought to be related to study drug. C. Other hemorrhagic events. | follow until Dec. 31, 2010
Number of ultrasounds and V/Q or CTA's required | follow until Dec. 31, 2010
Costs associated with each study arm, including that of drug, laboratory monitors, radiology procedures required, lengths of stay, and management of complications | follow until Dec. 31, 2010
Determine if negative D-D dimer can eliminate need for ultrasound analysis at follow-up visit. | follow until Dec. 31, 2010
Death due to any other cause than TED | follow until Dec. 31, 2010
Use of low molecular weight dextran | follow until Dec. 31, 2010
Use of nonsteroidal anti-inflammatory drugs | follow until Dec. 31, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Murray Bern, MD, Principal Investigator — New England Baptist Hospital
Locations (1):
- New England Baptist Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bern MM, Hazel D, Deeran E, Richmond JR, Ward DM, Spitz DJ, Mattingly DA, Bono JV, Berezin RH, Hou L, Miley GB, Bierbaum BE. Low dose compared to variable dose Warfarin and to Fondaparinux as prophylaxis for thromboembolism after elective hip or knee replacement surgery; a randomized, prospective study. Thromb J. 2015 Oct 7;13:32. doi: 10.1186/s12959-015-0062-0. eCollection 2015. PMID 26448724
- [Derived] Bern MM, Hazel D, Reilly DT, Adcock DM, Hou L. Effects of anticoagulation on markers of activation of clotting following major orthopedic surgery. Int J Lab Hematol. 2015 Oct;37(5):673-9. doi: 10.1111/ijlh.12384. Epub 2015 May 15. PMID 25975205